CLINICAL TRIAL: NCT07010536
Title: Effect of Immersive Virtual Reality-Based Music Therapy on Cognitive and Motor Skills in Subacute Stroke Patients
Brief Title: Effect of Virtual Reality-Based Music Therapy on Cognitive and Motor Skills in Subacute Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzan Aydın (Other)
Responsible Party: Sponsor-Investigator, Suzan Aydın, Principal Investigator, Physiotherapist, Lecturer and Ph.D. Candidate in Physical Therapy and Rehabilitation, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/020-1000
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Subacute Stroke; Virtual Reality; Immersive Virtual Reality; Cognitive Dysfunction; Motor Impairment
Keywords: Stroke; Music Therapy; Virtual Reality; Cognition Disorders; Motor Skills Disorders; Postural Balance
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Cognition Disorders; Motor Skills Disorders | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two parallel groups: a control group receiving only conventional physiotherapy, and an experimental group receiving conventional physiotherapy combined with immersive virtual reality-based music therapy. Both groups will receive interventions for 6 weeks, and outcomes will be compared between groups.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group allocation. Participants and care providers are not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy and Rehabilitation Group (Active Comparator): Participants in the control arm will receive conventional physiotherapy and rehabilitation exercises five days per week for six weeks, with sessions lasting approximately 60 minutes. The program includes:
  Strengthening exercises for upper and lower extremities
  Resistance training
  Aerobic exercises
  Basic and assisted parallel bar walking
  Skill courses on different surfaces
  Balance exercises on stable and unstable surfaces
  Static and dynamic balance training
  Fine motor skill exercises
  Weight transfer exercises aimed at improving postural stability
  Exercises will be tailored to individual patient capabilities and performed in various positions including standing, sitting, four-point kneeling, supine, and prone. The difficulty level will be adjusted based on patient performance and functional status.
  Interventions: Behavioral: Conventional Physiotherapy and Rehabilitation
- VR-Based Music Therapy Group (Experimental): Participants in the experimental arm will receive conventional physiotherapy and rehabilitation exercises five days per week for six weeks, each session lasting approximately 60 minutes. In addition to this, they will undergo immersive virtual reality (VR)-based music therapy sessions twice a week for 30 minutes per session over the same six-week period.
  The VR therapy is administered under the supervision of a licensed physiotherapist using the Oculus Quest 2 headset. The intervention includes three main components:
  Rhythm Exercises: Participants will engage in rhythm training by following clapping patterns streamed from the Brooklyn Music Factory YouTube channel, progressing from levels 1 to 4. During these exercises, participants clap their hands on a table to maintain the rhythm, which aims to improve motor coordination and timing.
  PianoVision Application: A virtual piano that utilizes hand-tracking technology to allow participants to play without physical controllers. The pian
  Interventions: Behavioral: VR-Based Music Therapy; Behavioral: Conventional Physiotherapy and Rehabilitation

INTERVENTIONS:
Behavioral: VR-Based Music Therapy — VR-Based Music Therapy Protocol:
  Participants undergo immersive VR sessions twice weekly for 6 weeks, each lasting 30 minutes, supervised by a physiotherapist. Each session includes three 10-minute activities with 2-minute breaks:
  Rhythm Exercises: Participants follow tempo by clapping on a table while watching Brooklyn Music Factory YouTube videos played within the VR headset (levels 1-4), progressing weekly.
  Ocean Rift: Exploration of calming underwater environments with marine life to enhance relaxation, attention, and cognition.
  PianoVision: Virtual piano exercises using hand tracking with the unaffected hand; difficulty increases from levels 0 to 4.
  Arms: VR-Based Music Therapy Group
Behavioral: Conventional Physiotherapy and Rehabilitation — Participants will receive conventional physiotherapy and rehabilitation exercises as follows:
  Upper and lower extremity strengthening exercises
  Resistance training exercises
  Aerobic exercises
  Basic and assisted parallel bar walking
  Skill courses on various surfaces
  Training on stable and unstable surfaces
  Static and dynamic balance exercises
  Fine motor skill exercises
  Weight transfer exercises to improve postural stability
  Exercises will be performed according to the patient's condition in standing, sitting, four-point kneeling, supine, and prone positions.
  Exercise difficulty will be adjusted based on the patient's performance and functional level.
  Sessions will be 60 minutes long, 5 days per week, for 6 weeks.

SUMMARY:
This clinical trial aims to investigate the effects of immersive virtual reality-based music therapy on cognitive and motor functions in individuals aged 50 to 75 years with subacute stroke (between 2 weeks and 6 months post-stroke). Participants will be randomly assigned to either a control group receiving conventional physiotherapy or an experimental group receiving conventional physiotherapy plus virtual reality-based music therapy.

The study will assess cognitive performance, upper extremity motor skills, stroke impact, balance, and spatial neglect before and after a 6-week intervention. All participants will be treated at Istanbul Aydın University VM Medical Park Hospital. The study has been approved by the ethics committee, and written informed consent will be obtained from all participants.

DETAILED DESCRIPTION:
This is a single-center, single bilind, randomized, controlled, prospective clinical trial designed to evaluate the effects of immersive virtual reality (VR)-based music therapy on cognitive functions, upper extremity motor skills, stroke impact, balance, and spatial neglect in patients with subacute stroke. The study targets individuals aged between 50 and 75 years who have experienced a stroke within the previous 2 weeks to 6 months. All participants will be recruited from Istanbul Aydın University VM Medical Park Hospital.

Participants will be stratified based on the side of hemispheric damage (right or left) and randomized into two equal groups (n=15 per group). The control group will receive conventional physiotherapy and rehabilitation 5 days per week for 6 weeks. The experimental group will receive the same conventional physiotherapy program along with additional immersive VR-based music therapy sessions twice a week. These VR sessions involve rhythm-based and music-supported tasks delivered through Oculus Quest 2 applications, including Ocean Rift and PianoVision.

Assessments will be performed at baseline and after the 6-week intervention period. Cognitive function will be assessed using standardized neuropsychological tools, and motor function will be evaluated through established stroke motor recovery scales. The Virtual Reality Sickness Questionnaire (VRSQ) will be administered after the first VR session to monitor adverse effects such as dizziness or nausea.

This trial adopts a stratified randomization method to enhance internal validity by balancing brain hemisphere involvement across groups. A power analysis conducted using G*Power (version 3.1) determined a sample size of 30 participants based on an effect size reported by Fan et al. (2024), with 95% power and α=0.05. The study protocol has been approved by the Non-Interventional Research Ethics Committee of Üsküdar University (Approval No: 61351342/020-1000, Date: March 27, 2025). Written informed consent will be obtained from all participants before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Age between 50 and 75 years
* Stroke onset more than 2 weeks and less than 6 months prior
* Diagnosis of unilateral hemiplegic stroke
* Preserved understanding, hearing, and speech abilities sufficient to engage with virtual reality games

Exclusion Criteria:

* Medically unstable condition
* Wheelchair use or inability to sit in a chair
* Cognitive impairment preventing comprehension of study procedures
* Hearing loss
* Severe visual impairment
* Refusal to participate in the study
* Epilepsy
* Migraine with aura
* History of motion sickness

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Global Cognitive Function as Assessed by the Montreal Cognitive Assessment (MoCA) at 6 Weeks | Baseline and 6 weeks after the start of intervention
  Cognitive function was assessed using the Montreal Cognitive Assessment (MoCA), a standardized screening tool for global cognitive functioning. The assessment was conducted face-to-face by a trained evaluator. The MoCA consists of tasks evaluating memory, attention, executive functions, language, visuospatial skills, abstraction, calculation, and orientation. Scores range from 0 to 30. Higher scores indicate better cognitive performance. A score of 26 or higher is generally considered normal.
Change from Baseline in Visual Memory as Assessed by the Benton Visual Retention Test - Form F at 6 Weeks | Baseline and 6 weeks after the intervention
  Visual memory was evaluated using the Benton Visual Retention Test (BVRT), Form F, a standardized neuropsychological test that assesses short-term visual memory, visual perception, and visuoconstructive skills. In this version, participants were shown 15 geometric designs, each for 10 seconds, and were instructed to reproduce each design from memory immediately after viewing. Each figure was scored based on established accuracy criteria. The outcome measure was the total number of correctly reproduced designs, with scores ranging from 0 to 15. Higher scores indicate better visual memory performance. Increased errors may reflect difficulties in memory, attention, or visual-spatial processing.
Change from Baseline in Working Memory Performance as Assessed by the Digit Span Test at 6 Weeks | Baseline and 6 weeks after the intervention
  Working memory was measured using the Digit Span subtest from the Wechsler Adult Intelligence Scale. The test consists of forward and backward repetition of digit sequences. Participants were asked to repeat sequences in the same order (forward) and reverse order (backward). Each correct sequence was scored, and the total score was recorded. Scores typically range from 0 to 30. Higher scores reflect greater working memory capacity.
Change from Baseline in Executive Function as Assessed by the Wisconsin Card Sorting Test (WCST) at 6 Weeks | Baseline and 6 weeks after the intervention
  Executive function was assessed using the Wisconsin Card Sorting Test (WCST), which evaluates cognitive flexibility and problem-solving. Participants were required to match cards based on undisclosed rules and adapt as the rules changed. The outcome measure is the number of correct categories completed. The maximum number of categories is 6. Higher scores reflect better executive functioning.
Change from Baseline in Upper Extremity Motor Function as Assessed by the Fugl-Meyer Assessment of Upper Extremity (FMA-UE) at 6 Weeks | Baseline and 6 weeks after the start of intervention
  Motor function of the upper limb will be assessed using the Fugl-Meyer Assessment of Upper Extremity (FMA-UE), a validated and widely used scale in stroke rehabilitation. The FMA-UE evaluates reflex activity, volitional movement within and out of synergy, grasp, coordination, and speed. Scores range from 0 to 66, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Change from Baseline in Balance Performance as Assessed by the Berg Balance Scale (BBS) at 6 Weeks | Baseline and 6 weeks after the start of intervention
  Balance performance will be assessed using the Berg Balance Scale (BBS), a validated tool to evaluate static and dynamic balance in individuals with stroke. The BBS consists of 14 tasks related to postural control and risk of falling. Each task is scored on a 5-point scale from 0 to 4, with a total score ranging from 0 to 56. Higher scores indicate better balance and lower risk of falls. Assessments will be conducted at baseline and 6 weeks post-intervention to evaluate changes in balance following immersive virtual reality-based music therapy.
Change from Baseline in Motor Recovery Assessed by Brunnstrom Staging at 6 Weeks | Baseline and 6 weeks after the start of intervention
  Brunnstrom Staging is used to evaluate motor recovery stages in stroke patients, assessing movement patterns and motor control progression. This measure will assess motor function improvements following immersive virtual reality-based music therapy. Assessments will be conducted at baseline and 6 weeks post-intervention.
Change from Baseline in Spatial Neglect Severity as Assessed by the Star Cancellation Test at 6 Weeks | Baseline and 6 weeks (only for participants with spatial neglect at baseline)
  Spatial neglect will be screened using the Star Cancellation Test (SCT), a validated subtest of the Behavioral Inattention Test (BIT). Participants are asked to cancel 54 small stars among distractor stimuli on a printed page. The total score is based on the number of correctly cancelled small stars. Scores range from 0 to 54, with scores of 43 or below indicating the presence of spatial neglect. Lower scores indicate more severe neglect. The test will be administered to all participants at baseline. Participants who score ≤43 will be considered to have spatial neglect, and for these individuals the test will be repeated at 6 weeks to evaluate change. Participants who do not meet the cutoff at baseline will not be retested.

OTHER OUTCOMES:
Virtual Reality Sickness Score After First Session as Assessed by the Virtual Reality Sickness Questionnaire (VRSQ) | After first VR session (Week 1)
  VR-induced sickness will be assessed using the Virtual Reality Sickness Questionnaire (VRSQ), a validated tool designed specifically for evaluating motion sickness symptoms in immersive virtual environments. The VRSQ includes 9 items categorized under two components: oculomotor symptoms (general discomfort, fatigue, eye strain, and difficulty focusing) and disorientation symptoms (headache, fullness in head, blurred vision, dizziness with eyes closed, and vertigo). Each item is scored on a 4-point Likert scale from 0 (none) to 3 (severe). Component scores are normalized to percentages and averaged to obtain the total score. Total scores range from 0 to 100, with higher scores indicating more severe VR sickness. The questionnaire will be administered immediately after the first VR session to evaluate tolerability and detect early side effects of immersive VR-based music therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Selen GÜR ÖZMEN, Associate Professor, Study Director — Bahçeşehir University
Locations (1):
- Istanbul Aydin University VM Medical Park Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all individual participant data (IPD) collected throughout the trial, including baseline characteristics, intervention details, outcome measures, and adverse events. The data will be de-identified to protect participant privacy and made available upon reasonable request to qualified researchers following publication of the main results.
Supporting Information: Study Protocol